CLINICAL TRIAL: NCT06473896
Title: Comparison of the Effect of Ketalar or Dexmedetomidine on Increased Sensitivity to Pain Induced Following Treatment With Remifentanil in Patients Undergoing a Laparoscopic Cholecystectomy
Brief Title: Effect of Ketalar or Dexmedetomidine on Increased Sensitivity to Pain Following Treatment With Remifentanil
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Zoya Haitov Ben Zikri, Manager of the anesthesia unit, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0173-23-ASF
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Cholecystectomy
MeSH Terms: interventions — Ketamine; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: The patients will be classified into 2 groups:
  The Ketalar group - who will receive, in addition to the general anesthesia, a bolus of Ketalar during induction and during the operation, continuous ketamine.
  The Dexmedetomidine group - in addition to the general anesthesia, they will also receive a Dexmedetomidine bolus in the induction and during the operation continuous Dexmedetomidine
Who Masked: Participant
Masking Description: The patients will not be exposed to the treatment arm they will receive
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketalar (Active Comparator): All patients will undergo general anesthesia using Fentanyl at a dose of 2 mcg/kg, Rocuronium at a dose of 0.6 mg/kg, Isoflurane during surgery and Remifentanil at a dose of 0.2-0.25 mcg/kg/min, 30 Minutes before the end of the operation, Morphine will be given at a dose of 0.1 mg/kg. Each patient will receive paracetamol during surgery.
  In addition to the general anesthesia, the patients in the Ketalar group will also receive a bolus of Ketalar at a dose of 0.3 mg/kg in induction + Propofol and Fentanyl and during the operation, continuous Ketalar at a dose of 5 mcg/kg/minute.
  Interventions: Drug: Ketalar
- Dexmedetomidine (Active Comparator): In addition to the general anesthesia, the patients in the Dexmedetomidine group will also receive a bolus of Ketalar at a dose of 0.3 mg/kg in induction + Propofol and Fentanyl and during the operation, continuous Ketalar at a dose of 5 mcg/kg/minute.
  In addition to the general anesthesia, the patients in the Dexmedetomidine group will also receive a bolus of Dexmedetomidine at a dose of 0.5 mg/kg for fifteen minutes + Propofol and Fentanyl, and during the operation, continuous Dexmedetomidine at a dose of 0.3 mcg/kg/hour.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Ketalar — a dissociative anesthetic used medically for induction and maintenance of anesthesia
  Other Names: Ketamine
  Arms: Ketalar
Drug: Dexmedetomidine — an agonist of α2-adrenergic receptors in certain parts of the brain used for sedation
  Other Names: Precedex
  Arms: Dexmedetomidine

SUMMARY:
Analgesia is one of the pillars of anesthesia. One of the common opiates for pain relief, with a short half-life, is Remifentanil. However, following Remifentanil treatment an increased sensitivity to pain [hyperalgesia] appears. The aim of the study is to compare the effects between complementary treatments, like Ketalar and Dexmedetomidine, in preventing increased sensitivity to pain after Remifentanil treatment

DETAILED DESCRIPTION:
Analgesia is one of the pillars of anesthesia. For many years, opiates were the basic ingredient in pain relief. The effectiveness of these substances in pain relief caused them to be overused which resulted in a global epidemic of addiction, morbidity and mortality due to the overuse of these drugs. Some of the options for realizing a reduction in the use of opiates include the use of drugs with a more predictable pharmacological profile and a short half-life, such as Remifentanil. This opiate is stronger than Morphine and its half-life remains within a few minutes, without accumulation even after prolonged infusion. Therefore, it seems that the use of remifentanil is ideal, especially for prolonged anesthesia.

One of the severe complications following treatment with Remifentanil is the appearance of increased sensitivity to pain [hyperalgesia] which results from a central sensitivity to pain and is expressed by stimulation of sensory receptors for pain in the nervous system (nociceptive sensitization). In order to alleviate the feeling of pain following the increased sensitivity to pain after treatment with opiates, as well as with Remifentanil, complementary treatments, such as Ketalar and dexmedetomidine, were offered. This study will compare the ability of Ketalar or Dexmedetomidine in alleviating increased sensitivity to pain after treatment with Remifentanil in patients who are candidates for laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

• Patients who are about to undergo alaparoscopic cholecystectomy under general anesthesia

Exclusion Criteria:

* Patients with sensitivity to the anesthetic
* Patients with chronic pain who are in regular treatment
* Urgent surgery
* Patients with ischemic heart disease
* Patients with known bradycardia
* Patients with a pacemaker
* Prolonged use of opiates
* Kidney/liver function problems

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Pain Level | Up to two hours after the end of the anesthesia process
  A record of pain level will be made using the Visual Analogue Scale. The score is determined by marking on 10-cm line between 0 - "no pain" to 10 - "the highest pain".
Pain killer consumption | Up to two hours after the end of the anesthesia process
  Treatment with morphine for pain relief

CONTACTS AND LOCATIONS:
Overall Officials: Sara Bar Yehuda, PhD, Study Director — Shamir (Asaf Harofe) medical center
Locations (1):
- Shamir (Asaf Harofe) Medical Center, Be’er Ya‘aqov, Israel

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be = will be provided as needed after receiving approval from the authorities of the Shamir (Asaf Harofe) medical center